CLINICAL TRIAL: NCT02788890
Title: Vital Signs Changes During Different Dental Procedures in Otherwise Healthy Adult Patients.
Brief Title: Vital Signs Changes During Dental Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Ra'ed Salma, Assistant Professor Oral and Maxillofacial Surgery, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: FRP/2016/43
Record Dates: First submitted 2016-05-23; First posted 2016-06-02 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Vital Signs Changes During Dental Procedures
MeSH Terms: interventions — Tooth Exfoliation

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The care provider was not aware of study objectives. The outcomes assessor was not involved in the data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (T0) (Active Comparator): The supragingival scaling without LA
  Interventions: Procedure: Scaling without LA
- Test Group 1 (T1) (Experimental): The simple restoration under LA
  Interventions: Procedure: Simple restoration under LA
- Test Group 2 (T2) (Experimental): The simple exodontia under LA
  Interventions: Procedure: Simple exodontia under LA

INTERVENTIONS:
Procedure: Scaling without LA — The patient will undergo a supragingival scaling procedure without local anesthesia
  Arms: Control Group (T0)
Procedure: Simple restoration under LA — The patient will undergo a simple dental restoration procedure under local anesthesia
  Arms: Test Group 1 (T1)
Procedure: Simple exodontia under LA — The patient will undergo a simple dental extraction procedure under local anesthesia
  Arms: Test Group 2 (T2)

SUMMARY:
The study will evaluate the vital signs changes during 3 different dental procedures performed for the same patient by the same dentist. The patients will be selected randomly and should all be healthy adults.

The aim is to look for any significant changes in the major vital signs (heart rate, respiratory rate, blood pressure, peripheral capillary oxygen saturation (SpO2) and body temperature) during specified dental procedures (scaling, simple restoration, and simple exodontia) and compare the changes between the 3 procedures.

ELIGIBILITY:
Inclusion Criteria:

* The patients included are the ones planned for the following 3 dental treatments in 3 separate visits to done by the same dentist: supragingival scaling without local anesthesia (LA), simple dental extraction under LA, and simple restoration under LA.

Exclusion Criteria:

* Patients under 18 years old
* Patients with a known medical history of any systemic disease like hypertension, diabetes, and bleeding disorders
* Patients with history of cardiac surgery; including pace maker insertion
* Patients on medications
* Smokers, alcoholics, and drug abusers
* Pregnant patients
* Patients with an acute infection with or without fever
* Patients with a preoperative pain score of 4 or more on a visual analogue scale out of 10; where 0 = no pain and 10 = worst pain imaginable
* Patients with 2 or more simultaneous dental procedures per visit
* Patients with undiagnosed hypertension who are found to be hypertensive according to the World Health Organization (WHO) definition on the base-line preoperative readings

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Change in Body Temperature (BT) during Periodontal Therapy from the baseline BT | Baseline, intraoperative, 5-min postoperative
  Body temperature measured in Celsius using infrared non-contact digital thermometer
Change in Body Temperature (BT) during Operative Procedure from the baseline BT | Baseline, during anesthesia injection, intraoperative, 5-min postoperative
  Body temperature measured in Celsius using infrared non-contact digital thermometer
Change from baseline Body Temperature (BT) during Dental Extraction from the baseline BT | Baseline, during anesthesia injection, intraoperative, 5-min postoperative
  Body temperature measured in Celsius using infrared non-contact digital thermometer
Change in Respiratory Rate (RR) during Periodontal Therapy from the baseline RR | Baseline, intraoperative, 5-min postoperative
  Respiratory rate is measured by observing the chest and/or abdominal movements and count the number of respirations out loud for one full minute. One respiration consists of one complete rise and fall of the chest (inhalation and exhalation of air)
Change in Respiratory Rate (RR) during Operative Procedure from the baseline RR | Baseline, during anesthesia injection, intraoperative, 5-min postoperative
  Respiratory rate is measured by observing the chest and/or abdominal movements and count the number of respirations out loud for one full minute. One respiration consists of one complete rise and fall of the chest (inhalation and exhalation of air)
Change in Respiratory Rate (RR) during Dental Extraction from the baseline RR | Baseline, during anesthesia injection, intraoperative, 5-min postoperative
  Respiratory rate is measured by observing the chest and/or abdominal movements and count the number of respirations out loud for one full minute. One respiration consists of one complete rise and fall of the chest (inhalation and exhalation of air)
Change in Heart Rate (HR) during Periodontal Therapy from the baseline HR | Baseline, intraoperative, 5-min postoperative
  The heart rate will be recorded using a non-invasive infrared pulse oximeter placed on the patient's left index finger attached to an ambulatory digital monitor
Change in Heart Rate (HR) during Operative Procedure from the baseline HR | Baseline, during anesthesia injection, intraoperative, 5-min postoperative
  The heart rate will be recorded using a non-invasive infrared pulse oximeter placed on the patient's left index finger attached to an ambulatory digital monitor
Change in Heart Rate (HR) during Dental Extraction from the baseline HR | Baseline, during anesthesia injection, intraoperative, 5-min postoperative
  The heart rate will be recorded using a non-invasive infrared pulse oximeter placed on the patient's left index finger attached to an ambulatory digital monitor
Change in Peripheral Oxygen Saturation (SpO2) during Periodontal Therapy from the baseline SpO2 | Baseline, intraoperative, 5-min postoperative
  The SpO2 will be recorded using a non-invasive infrared pulse oximeter placed on the patient's index finger attached to an ambulatory digital monitor
Change in Peripheral Oxygen Saturation (SpO2) during Operative Procedure from the baseline SpO2 | Baseline, during anesthesia injection, intraoperative, 5-min postoperative
  The SpO2 will be recorded using a non-invasive infrared pulse oximeter placed on the patient's index finger attached to an ambulatory digital monitor
Change in Peripheral Oxygen Saturation (SpO2) during Dental Extraction from the baseline SpO2 | Baseline, during anesthesia injection, intraoperative, 5-min postoperative
  The SpO2 will be recorded using a non-invasive infrared pulse oximeter placed on the patient's index finger attached to an ambulatory digital monitor
Change in Systolic Blood Pressure (SBP) during Periodontal Therapy from the baseline SBP | Baseline, intraoperative, 5-min postoperative
  The blood pressure BP will be measured utilizing the NIBP (noninvasive blood pressure) measurement tool attached to an ambulatory digital monitor and recorded in mmHg
Change in Systolic Blood Pressure (SBP) during Operative Procedure from the baseline SBP | Baseline, during anesthesia injection, intraoperative, 5-min postoperative
  The blood pressure BP will be measured utilizing the NIBP (noninvasive blood pressure) measurement tool attached to an ambulatory digital monitor and recorded in mmHg
Change in Systolic Blood Pressure (SBP) during Dental Extraction from the baseline SBP | Baseline, during anesthesia injection, intraoperative, 5-min postoperative
  The blood pressure BP will be measured utilizing the NIBP (noninvasive blood pressure) measurement tool attached to an ambulatory digital monitor and recorded in mmHg
Change in Diastolic Blood Pressure (DBP) during Periodontal Therapy from the baseline DBP | Baseline, intraoperative, 5-min postoperative
  The blood pressure BP will be measured utilizing the NIBP (noninvasive blood pressure) measurement tool attached to an ambulatory digital monitor and recorded in mmHg MAP= (Systolic BP + 2*Diastolic BP)/3 And recorded in mmHg
Change in Diastolic Blood Pressure (DBP) during Operative Procedure from the baseline DBP | Baseline, during anesthesia injection, intraoperative, 5-min postoperative
  The blood pressure BP will be measured utilizing the NIBP (noninvasive blood pressure) measurement tool attached to an ambulatory digital monitor and recorded in mmHg
Change in Diastolic Blood Pressure (DBP) during Dental Extraction from the baseline DBP | Baseline, during anesthesia injection, intraoperative, 5-min postoperative
  The blood pressure BP will be measured utilizing the NIBP (noninvasive blood pressure) measurement tool attached to an ambulatory digital monitor and recorded in mmHg

SECONDARY OUTCOMES:
Change in Pulse Pressure (PP) during Periodontal Therapy from the baseline PP | Baseline, intraoperative, 5-min postoperative
  The blood pressure BP will be measured utilizing the NIBP (noninvasive blood pressure) measurement tool attached to an ambulatory digital monitor. The PP is then calculated as the systolic and diastolic blood pressure difference and recorded in mmHg
Change in Pulse Pressure (PP) during Operative Procedure from the baseline PP | Baseline, during anesthesia injection, intraoperative, 5-min postoperative
  The blood pressure BP will be measured utilizing the NIBP (noninvasive blood pressure) measurement tool attached to an ambulatory digital monitor. The PP is then calculated as the systolic and diastolic blood pressure difference and recorded in mmHg
Change in Pulse Pressure (PP) during Dental Extraction from the baseline PP | Baseline, during anesthesia injection, intraoperative, 5-min postoperative
  The blood pressure BP will be measured utilizing the NIBP (noninvasive blood pressure) measurement tool attached to an ambulatory digital monitor. The PP is then calculated as the systolic and diastolic blood pressure difference and recorded in mmHg
Change in Mean Arterial Pressure (MAP) during Periodontal Therapy from the baseline MAP | Baseline, intraoperative, 5-min postoperative
  The blood pressure BP will be measured utilizing the NIBP (noninvasive blood pressure) measurement tool attached to an ambulatory digital monitor. The MAP is then calculated using the following equation:
  MAP= (Systolic BP + 2*Diastolic BP)/3 And recorded in mmHg
Change in Mean Arterial Pressure (MAP) during Operative Procedure from the baseline MAP | Baseline, during anesthesia injection, intraoperative, 5-min postoperative
  The blood pressure BP will be measured utilizing the NIBP (noninvasive blood pressure) measurement tool attached to an ambulatory digital monitor. The MAP is then calculated using the following equation:
  MAP= (Systolic BP + 2*Diastolic BP)/3 And recorded in mmHg
Change in Mean Arterial Pressure (MAP) during Dental Extraction from the baseline MAP | Baseline, during anesthesia injection, intraoperative, 5-min postoperative
  The blood pressure BP will be measured utilizing the NIBP (noninvasive blood pressure) measurement tool attached to an ambulatory digital monitor. The MAP is then calculated using the following equation:
  MAP= (Systolic BP + 2*Diastolic BP)/3 And recorded in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Ra'ed G Salma, Principal Investigator — Riyadh Colleges of Dentistry and Pharmacy
Locations (1):
- Riyadh Colleges of Dentistry & Pharmacy, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided